CLINICAL TRIAL: NCT07080255
Title: Tight-Rope Augmented Adams Berger Reconstruction Improves Outcome in Chronic Distal Radioulnar Joint İnstability: A Prospective Randomized Trial
Brief Title: Tight-Rope Augmented Adams Berger Technique for Distal Radioulnar Joint Instability
Acronym: Druj Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Bulent KARSLIOGLU, Associate Professor, Orthopedic Surgeon, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Druj Instability Surgery
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Distal Radioulnar Joint Instability; Chronic Post-Traumatic DRUJ Instability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adams-Berger Reconstruction Only (Active Comparator): Patients in this arm underwent anatomical reconstruction of the distal radioulnar joint (DRUJ) using the standard Adams-Berger technique. A palmaris longus tendon graft was harvested and passed through bone tunnels in the radius and ulna to reconstruct both palmar and dorsal radioulnar ligaments. No additional device was used.
  Interventions: Procedure: Adams-Berger Reconstruction
- Adams-Berger Reconstruction with TightRope® Augmentation (Experimental): In addition to the Adams-Berger anatomical ligament reconstruction, this group received TightRope® (Double Loop Lift System) augmentation for added dynamic stabilization. A suture-button construct was applied across the radius and ulna to enhance joint stability and allow early mobilization.
  Interventions: Device: TightRope®-Augmented Adams-Berger Reconstruction

INTERVENTIONS:
Procedure: Adams-Berger Reconstruction — The Adams-Berger procedure involves anatomical reconstruction of the distal radioulnar joint (DRUJ) ligaments using a palmaris longus tendon graft. Bone tunnels are drilled in the radius and ulna, and the graft is passed through these tunnels to reconstruct the dorsal and palmar radioulnar ligaments. This technique is designed to restore stability in patients with chronic post-traumatic DRUJ instability.
  Other Names: Anatomical DRUJ ligament reconstruction
  Arms: Adams-Berger Reconstruction Only
Device: TightRope®-Augmented Adams-Berger Reconstruction — This intervention combines the standard Adams-Berger procedure with the addition of the TightRope® (Double Loop Lift System) device to provide dynamic stabilization of the DRUJ. The TightRope® system consists of a FiberWire suture passed through 2.7 mm bone tunnels in the radius and ulna and secured with cortical metal buttons. It allows for early mobilization and enhanced postoperative joint stability.
  Other Names: TightRope®, Double Loop Lift System
  Arms: Adams-Berger Reconstruction with TightRope® Augmentation

SUMMARY:
Brief Summary This clinical study evaluated a new surgical technique for treating chronic instability of the distal radioulnar joint (DRUJ), a joint in the wrist responsible for forearm rotation. Chronic DRUJ instability, often resulting from trauma, may lead to wrist pain, weakness, and restricted movement. One established surgical intervention is the Adams-Berger procedure, which reconstructs DRUJ ligaments using a tendon graft.

This investigation aimed to enhance the traditional Adams-Berger procedure by incorporating a suture-button system, TightRope®, which offers dynamic stabilization. TightRope® is a non-absorbable suture construct fixed between the radius and ulna to provide semi-rigid support, potentially facilitating earlier mobilization and improved healing.

Between January 2015 and January 2020, 36 adult patients with chronic post-traumatic DRUJ instability unresponsive to six months of conservative treatment were enrolled in a randomized controlled trial. Patients were randomly assigned to either undergo the standard Adams-Berger procedure (Group A) or the same procedure with additional TightRope® stabilization (Group B). All surgeries were conducted by a single orthopedic surgeon, with informed consent obtained preoperatively.

Outcomes were assessed at 3 and 6 months postoperatively using standardized measures of function, pain, grip strength, and range of motion. Results demonstrated superior improvements in grip strength, pain reduction, and functional recovery in the TightRope® group. Notably, no cases of recurrent instability occurred in Group B, while two cases were observed in Group A.

These findings suggest that TightRope® augmentation of the Adams-Berger procedure offers improved stabilization and expedited functional recovery, representing a promising advancement in the surgical treatment of DRUJ instability.

DETAILED DESCRIPTION:
Detailed Description (Revised) Chronic distal radioulnar joint (DRUJ) instability is a disabling condition that compromises wrist function and quality of life. It typically arises from trauma and may persist despite extended conservative management. The DRUJ comprises complex bony and soft tissue components, with the triangular fibrocartilage complex (TFCC) being critical to stability. When the TFCC is irreparably damaged, surgical reconstruction is often indicated.

The Adams-Berger procedure, an anatomical reconstruction technique, is commonly utilized to restore dorsal and palmar radioulnar ligaments using a tendon graft. While this method has demonstrated clinical efficacy, limitations include residual instability and delayed functional recovery. To address these challenges, a modified surgical technique integrating the TightRope® suture-button system into the Adams-Berger procedure was developed, aiming to enhance biomechanical stability.

This prospective, randomized controlled trial was conducted between January 2015 and January 2020. Thirty-six adult patients with post-traumatic, dynamic DRUJ instability and a minimum of six months of failed conservative management were enrolled. Randomization into two groups was performed using sealed opaque envelopes: Group A received the standard Adams-Berger procedure, while Group B underwent the same procedure with additional TightRope® augmentation.

All surgical procedures were performed by a single orthopedic surgeon. In both groups, the palmaris longus tendon was harvested and used to reconstruct the dorsal and palmar distal radioulnar ligaments. For Group B, an additional 2.7 mm bone tunnel was drilled through the distal radius and ulna, and the TightRope® device was positioned and tensioned with the forearm in a neutral position. Fluoroscopic confirmation of placement was obtained intraoperatively.

Postoperative management included a three-week period of long-arm splinting, followed by passive-assisted motion and progressive strengthening exercises. Functional outcomes, pain, grip strength, range of motion, and DRUJ stability were evaluated at baseline, 3 months, and 6 months postoperatively. Assessment tools included the QuickDASH questionnaire, visual analog scale (VAS) for pain, dynamometric grip strength testing, and clinical examination of pronation-supination arc and joint stability.

Both groups showed significant improvements in functional and pain outcomes. However, Group B (TightRope®-augmented) demonstrated statistically superior results in QuickDASH scores, grip strength, and range of motion. Recurrent instability was observed in two patients in Group A, whereas no recurrence was noted in Group B.

Advantages of the TightRope®-augmented technique include:

Dynamic stabilization without the need for hardware removal

Early initiation of mobilization due to semi-rigid fixation

Decreased risk of recurrent instability

Simplified intraoperative application using fluoroscopic guidance

Study limitations include a relatively short follow-up duration and the necessity for further investigation into optimal

ELIGIBILITY:
Inclusion Criteria:

Male patients aged between 18 and 47 years

Clinical diagnosis of chronic post-traumatic distal radioulnar joint (DRUJ) instability

Persistent ulnar-sided wrist pain refractory to at least 6 months of conservative treatment

Intraoperative confirmation of irreparable triangular fibrocartilage complex (TFCC) injury

Intact articular surfaces of the distal radius and ulna

Adequate palmar or dorsal rim of the sigmoid notch confirmed radiologically

Willingness to participate and ability to provide informed consent

Exclusion Criteria:

Evidence of DRUJ arthritis on imaging

Ulnar impaction syndrome

Extensor carpi ulnaris (ECU) tendon subluxation or tear

Inadequate sigmoid notch morphology (palmar/dorsal rim deficiency)

Age <18 or >47 years

Previous surgery on the affected wrist

Neurological or systemic conditions affecting wrist function

Patients unwilling or unable to comply with follow-up protocol

Ages: 18 Years to 47 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Change in QuickDASH Score from Baseline to 6 Months Postoperatively | Baseline and 6 Months Postoperative
  The Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) score is a validated patient-reported outcome measure used to assess upper extremity function. The scale ranges from 0 to 100, with lower scores indicating better functional status and less disability. The change in QuickDASH score from the preoperative baseline to the 6-month postoperative follow-up will be used to evaluate the degree of functional improvement after surgery.

SECONDARY OUTCOMES:
Change in Visual Analog Scale (VAS) Score from Baseline to 3 Months | Baseline and 3 Months Postoperative
  Pain intensity was assessed using the Visual Analog Scale (VAS), a validated 10-point scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Higher scores represent greater pain intensity. Changes in VAS scores from the preoperative baseline to the 3-month postoperative period were recorded to evaluate pain reduction.
Change in Hand Grip Strength from Baseline to 6 Months | Baseline and 6 Months Postoperative
  Grip strength was measured in kilograms using a calibrated hand-held dynamometer, with the participant's elbow positioned at 90° flexion. Three consecutive trials were performed, and the average value (in kg) was recorded. The change in grip strength from the preoperative baseline to the 6-month postoperative follow-up was assessed to evaluate functional recovery.
Limitation in Pronation-Supination Range of Motion at 6 Months | 6 Months Postoperative
  The range of forearm rotation, including pronation and supination, was measured clinically using a goniometer during physical examination. Measurements were recorded in degrees. Any limitation in motion was documented at the 6-month postoperative visit to assess residual functional deficits.
Recurrence of Distal Radioulnar Joint Instability at 6 Months | 6 Months Postoperative
  Recurrent distal radioulnar joint (DRUJ) instability was assessed clinically during postoperative follow-up visits using physical examination techniques, including evaluation for painful clunking, increased translation, and patient-reported discomfort. Instability was classified as either present or absent at the 6-month postoperative evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Cemil Tascioglu Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No